CLINICAL TRIAL: NCT04392440
Title: Pilot Testing of a Communication Intervention to Promote Shared Dialysis Decision Making in Older Patients With Chronic Kidney Disease (DIAL-SDM Trial)
Brief Title: Shared Decision Making in Dialysis
Acronym: DIAL-SDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Fahad Saeed, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00004907; K23DK121939 (NIH)
Record Dates: First submitted 2020-05-01; First posted 2020-05-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: End Stage Renal Disease; Chronic Kidney Diseases
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental)
  Interventions: Behavioral: DIAL-SDM
- control (Other): Usual care
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: DIAL-SDM — Communication intervention for nephrologists and coaching intervention for patients.
  Arms: intervention
Other: usual care — regular nephrology care
  Arms: control

SUMMARY:
Older patients ≥65 years with chronic kidney disease (CKD) face challenges in decision making about dialysis. These patients report little effort by physicians to elicit treatment preferences, discuss prognoses, or explain the burdens/benefits of dialysis options including conservative management. Older patients with CKD often prefer maintaining the quality of life over prolonging life, and many regret their decision to start dialysis: nearly one quarter withdraw from dialysis each year. Shared dialysis decision-making requires active engagement between nephrologists and patients to align patient, caregiver, and physician communication around common goals. The proposed study is a pilot randomized cluster trial of a dialysis shared decision-making (DIAL-SDM) intervention for nephrologists (n=20) and their patients ≥65 years old (n=60) with an estimated glomerular filtration rate (eGFR) of ≤ 20 ml/min/ /1.73 m2. Nephrologists in the Intervention Group will receive 3 communication training sessions, delivered by a standardized patient instructor (SPI) who enact clinical scenarios and offer feedback. In parallel, patients (and caregivers, if available) will receive 2 coaching sessions provided by health coaches, who will explore each patient's relevant contextual information (values, preferences, and goals), and help them identify and practice important questions for their nephrologist. Nephrologists in the Control Group will provide their patients with usual care. The study outcomes will be assessed during two nephrology office visits and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

For nephrologist:

* Member of Strong nephrology group working at Strong Memorial Hospital
* Treat patients with CKD

For patients:

* Age ≥65 years old
* Presence of advanced CKD stage 4 or 5 (i.e. e GFR ≤ 20 ml/min)
* Patient's nephrologist is enrolled in the study, and has seen that nephrologist at least once
* Speaks English
* Have not attended a dialysis education class or met with the dialysis education coordinator.
* Have not made a dialysis decision

For Caregivers:

* Self-identified caregiver (per definition:"family member, partner, friend or someone else who is involved with your health care issues, for example, someone who you talk to about personal issues including medical decisions or who comes to doctor appointments with you. This person may also help with routine day-to-day activities, like transportation or paperwork.")
* 21 years of age or older.

Exclusion Criteria:

For Nephrologists:

- Expecting to leave in six months.

For Patients:

* Patient has already been seen by a palliative care clinician or is enrolled in hospice
* Is already on dialysis
* Hospitalized at the time of recruitment
* Cognitive impairment
* Does not speak English

For Caregivers:

* If Support is offered primarily in a professional role (e.g., clergy).
* Cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
feasibility of DIAL-SDM intervention | Approximately 12 months
  This outcome will be measured in 30 patients in the Intervention Group
acceptability of DIAL-SDM intervention | Approximately 12 months
  This outcome will be measure in 30 patients in the Intervention Group
fidelity of DIAL-SDM intervention | Approximately 12 months
  This outcome will be measured by looking at the fidelity in which the interventionists complete the intervention checklist after each visit for 30 patients in the Intervention Group.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes